CLINICAL TRIAL: NCT04337515
Title: A Feasibility Study of Using the CiniMacs® Device for Alpha/Best T-Cell Depletion in Stem Cell Transplant Recipients
Brief Title: A Feasibility Study Using CLINIMACS® for Alpha/Beta T-Cell Depletion in Stem Cell Transplant
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Christopher Dvorak (Other)
Responsible Party: Sponsor-Investigator, Christopher Dvorak, Professor of Pediatrics, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-28063
Record Dates: First submitted 2020-02-27; First posted 2020-04-07 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Graft Vs Host Disease; Graft-versus-host-disease
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Patients receiving allogeneic hematopoietic cell transplant (Experimental): The test product is a stem cell product which has been alpha-beta T- cell depleted using the CliniMACS system. Alpha-beta T-cell depleted cells are given intravenously over a period of time as dictated by the final volume of the infused product (5 ml/kg/hour).
  The target dose of CD34+ cells is ≥20x10^6/kg, but a minimum of
  ≥2.5x10^6/kg is required. The target dose of T-cell receptor (TCR) alpha-beta CD3+ cells is ≤1x10^5/kg.
  Interventions: Device: CliniMacs®

INTERVENTIONS:
Device: CliniMacs® — CliniMACS® CD34 Reagent System is now indicated for processing hematopoietic progenitor cells collected by apheresis (PBSC) from an allogeneic, HLA-identical MSD to obtain a CD34+ cell-enriched population for hematopoietic reconstitution following a myeloablative preparative regimen without the need for additional GVHD prophylaxis in patients with AML in first morphologic complete remission (CR1).
  Other Names: CliniMACS® CD34 Reagent System

SUMMARY:
Patients in need of an allogeneic hematopoietic cell transplant (HCT) are at risk of developing graft-versus-host-disease (GVHD). In certain clinical situations, the optimal approach to minimize the risk of GVHD is to perform ex vivo alpha-beta T-cell depletion of the donor cells. However, the CliniMACS® Device is FDA-approved only for a narrow indication. All other uses of ex vivo processed cells must be done under a feasibility study protocol.

DETAILED DESCRIPTION:
The original CliniMACS® device (CD34 Reagent System) employs a reagent consisting of an antibody that specifically binds to blood cells that express the CD34+ surface marker (hematopoietic stem cells or blood stem cells). The CD34 antibody is conjugated to an iron-containing particle that is only nanometers in size and safe for infusion. The enrichment of CD34+ cells is accomplished by passing the antibody/magnetically-labeled cell suspension through a magnetic separation column, which is provided as part of a single-use disposable tubing set. Magnetically-labeled CD34+ target cells are retained within the separation column, while the unlabeled cells flow through. Recovery of CD34+ cells is achieved by removing the magnetic field and eluting the targeted CD34+ stem cells into a collection bag.

On January 24, 2014, the FDA approved the CliniMACS CD34 Reagent System as a Humanitarian Use Device for the prevention of graft-versus-host disease (GVHD) in patients with acute myeloid leukemia (AML) in first complete remission undergoing allogeneic HCT from a matched related donor. Humanitarian Use Device (HUD) is a device that is intended to benefit patients by treating or diagnosing a disease or condition that affects or is manifested in fewer than 4,000 individuals in the United States per year. The CliniMACS® CD34 Reagent System is now indicated for processing hematopoietic progenitor cells collected by apheresis (PBSC) from an allogeneic, Human Leukocyte Antigen (HLA)-identical matched sibling donor (MSD) to obtain a CD34+ cell-enriched population for hematopoietic reconstitution following a myeloablative preparative regimen without the need for additional GVHD prophylaxis in patients with AML in first morphologic complete remission (CR1). The approval as an HUD, however, asserts that there was sufficient information for the FDA to determine that the device does not pose an unreasonable or significant risk of illness or injury. Furthermore, the clinical data supported the premise of a "probable benefit"; in that the risk to health outweighs the risk of injury or illness from its use, taking into account the probable risks and benefits of currently available devices or alternative forms of treatment.19 The CliniMACS CD34 Reagent System was shown to meet these requirements.

Uses of the CliniMACS CD34 Reagent System beyond MSD PBSC HCT for AML in CR1 are currently not FDA approved and therefore considered research, even though CD34-selection is widely considered to be a standard-of-care option for haploidentical HCT. In Europe, the European Medicines Agency (EMA) has made the CliniMACs System components available as Conformité Européene (CE) marked medical devices, and "any clinical application of the target cells is exclusively within the responsibility of the user of a CliniMACS System."

The CD34-selection system has been widely used in haploidentical HCTs, with the first patient treated at University of California, San Francisco (UCSF) in 2002. Since then, CD34-selection has facilitated over 70 HCTs at UCSF on 2 successive protocols (#01151 and #10082). However, the removal of almost all cells beyond those which are CD34+ leads to minimal passive transfer of immunity. It is therefore complicated by a slow recovery of immunity, with high rates of life-threatening viral infections, and an appreciable degree of transplant-related mortality (TRM).

Beginning in 2014, a new approach to ex vivo processing of stem cells was developed with a goal of mainly replacing the older CD34-selection technology. This technique utilizes negative depletion of the cells thought to be most responsible for the development of aGVHD, the alpha-beta T-cell Receptor positive T-cells.

All trials of alpha-beta T-cell depleted have included simultaneous depletion of CD19+ B cells from the donor graft. All references to "alpha-beta T-cell depletion" herein implies simultaneous Cluster of Differentiation antigen (CD)19+ depletion as well.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 0-30 years of age at time of transplant admission
* Documentation of a disease requiring HCT
* A donor (mismatched related or unrelated) must be located who are healthy and willing, and whom are able to donate bone marrow (BM) or peripheral blood stem cells (PBSC). Matched related donors may be used for patients with Fanconi Anemia.
* Written informed consent (and assent when applicable) obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study

Exclusion Criteria:

* Pregnant, breastfeeding, or unwilling to practice birth control during participation in the study
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data
* Presence of a healthy and willing HLA-identical related donor (except when the patient has Fanconi Anemia).
* Patient with an anticipated life expectancy of <1 month
* Patients with known hypersensitivity to murine (mouse) proteins or iron dextran

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-12-19 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2035-01-01 (Estimated)

PRIMARY OUTCOMES:
100-day incidence of Grade III-IV acute GVHD | 100 days
  The cumulative incidence of Grade III-IV acute GVHD at Day 100 will be summarized by incidence curves. GVHD evaluations will be performed using standard criteria.37 Patients with graft rejection will be censored.

SECONDARY OUTCOMES:
30-day incidence of engraftment | 30 days
  The cumulative incidence of donor cell engraftment at 30 days will be summarized by incidence curves. Engraftment will be defined as ANC recovery (>500 x 3 days) with evidence of donor myeloid cells on chimerism analysis, OR, for non-myeloablative HCTs, evidence of donor cells on chimerism analysis.
1-year incidence of transplant-related mortality | 12 months
  The cumulative incidence of transplant-related mortality at 1-year will be summarized by incidence curves.
1-year incidence of systemic steroid-requiring chronic GVHD | 12 months
  The cumulative incidence of systemic steroid-requiring chronic GVHD at 1-year will be summarized by incidence curves. GVHD evaluations will be performed using standard criteria.
1-year incidence of autoimmunity requiring intervention with immunosuppressive agents as treatment. | 12 months
  The cumulative incidence of autoimmunity at 1-year will be summarized by incidence curves
180-day incidence of T-cell reconstitution (CD4+ T-cell count >200 and proliferation to PHA >50% control). | 180 days
  The incidence of T-cell reconstitution at Day 180 will be summarized by numbers and percentages of subjects in corresponding categories. T cell reconstitution is defined as a CD4+ T-cell count >200 and Proliferation to PHA >50% control

CONTACTS AND LOCATIONS:
Overall Officials: Christopher C Dvorak, MD, Principal Investigator — Professor of Clinical Pediatrics
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leung W, Campana D, Yang J, Pei D, Coustan-Smith E, Gan K, Rubnitz JE, Sandlund JT, Ribeiro RC, Srinivasan A, Hartford C, Triplett BM, Dallas M, Pillai A, Handgretinger R, Laver JH, Pui CH. High success rate of hematopoietic cell transplantation regardless of donor source in children with very high-risk leukemia. Blood. 2011 Jul 14;118(2):223-30. doi: 10.1182/blood-2011-01-333070. Epub 2011 May 25. PMID 21613256
- [Background] Klein OR, Buddenbaum J, Tucker N, Chen AR, Gamper CJ, Loeb D, Zambidis E, Llosa NJ, Huo JS, Robey N, Holuba MJ, Kasamon YL, McCurdy SR, Ambinder R, Bolanos-Meade J, Luznik L, Fuchs EJ, Jones RJ, Cooke KR, Symons HJ. Nonmyeloablative Haploidentical Bone Marrow Transplantation with Post-Transplantation Cyclophosphamide for Pediatric and Young Adult Patients with High-Risk Hematologic Malignancies. Biol Blood Marrow Transplant. 2017 Feb;23(2):325-332. doi: 10.1016/j.bbmt.2016.11.016. Epub 2016 Nov 22. PMID 27888014
- [Background] Berger M, Lanino E, Cesaro S, Zecca M, Vassallo E, Faraci M, De Bortoli M, Barat V, Prete A, Fagioli F. Feasibility and Outcome of Haploidentical Hematopoietic Stem Cell Transplantation with Post-Transplant High-Dose Cyclophosphamide for Children and Adolescents with Hematologic Malignancies: An AIEOP-GITMO Retrospective Multicenter Study. Biol Blood Marrow Transplant. 2016 May;22(5):902-9. doi: 10.1016/j.bbmt.2016.02.002. Epub 2016 Feb 6. PMID 26860636
- [Background] Abboud R, Keller J, Slade M, DiPersio JF, Westervelt P, Rettig MP, Meier S, Fehniger TA, Abboud CN, Uy GL, Vij R, Trinkaus KM, Schroeder MA, Romee R. Severe Cytokine-Release Syndrome after T Cell-Replete Peripheral Blood Haploidentical Donor Transplantation Is Associated with Poor Survival and Anti-IL-6 Therapy Is Safe and Well Tolerated. Biol Blood Marrow Transplant. 2016 Oct;22(10):1851-1860. doi: 10.1016/j.bbmt.2016.06.010. Epub 2016 Jun 16. PMID 27318038
- [Background] Handgretinger R, Klingebiel T, Lang P, Schumm M, Neu S, Geiselhart A, Bader P, Schlegel PG, Greil J, Stachel D, Herzog RJ, Niethammer D. Megadose transplantation of purified peripheral blood CD34(+) progenitor cells from HLA-mismatched parental donors in children. Bone Marrow Transplant. 2001 Apr;27(8):777-83. doi: 10.1038/sj.bmt.1702996. PMID 11477433
- [Background] Mancusi A, Ruggeri L, Velardi A. Haploidentical hematopoietic transplantation for the cure of leukemia: from its biology to clinical translation. Blood. 2016 Dec 8;128(23):2616-2623. doi: 10.1182/blood-2016-07-730564. Epub 2016 Oct 3. PMID 27697774
- [Background] Ortin M, Raj R, Kinning E, Williams M, Darbyshire PJ. Partially matched related donor peripheral blood progenitor cell transplantation in paediatric patients adding fludarabine and anti-lymphocyte gamma-globulin. Bone Marrow Transplant. 2002 Sep;30(6):359-66. doi: 10.1038/sj.bmt.1703667. PMID 12235520
- [Derived] Dvorak CC, Long-Boyle JR, Holbrook-Brown L, Abdel-Azim H, Bertaina A, Vatsayan A, Talano JA, Bunin N, Anderson E, Flower A, Lalefar N, Higham CS, Kapoor N, Klein O, Odinakachukwu MC, Cho S, Jacobsohn DA, Collier W, Pulsipher MA. Effect of rabbit ATG PK on outcomes after TCR-alphabeta/CD19-depleted pediatric haploidentical HCT for hematologic malignancy. Blood Adv. 2024 Dec 10;8(23):6003-6014. doi: 10.1182/bloodadvances.2024012670. PMID 39042892